CLINICAL TRIAL: NCT03796988
Title: Autologous Regeneration of Tissue (ART) for Wound Healing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: Medline Industries (Industry)
Responsible Party: Principal Investigator, Hadar Lev-Tov, Assistant Professor, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20180154
Record Dates: First submitted 2019-01-03; First posted 2019-01-08 (Actual); Results first posted 2025-04-23 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Wound of Skin
Keywords: Chronic Wound
MeSH Terms: interventions — Reproductive Techniques, Assisted

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Intervention arm (Experimental): The donor area will be anesthetized with injected local anesthesia, harvested with the ART device, and bandaged with an occlusive dressing. The skin harvested will be placed on the recipient wound area. The area will be bandaged will a non-stick silicone dressing (covered by appropriate primary and secondary dressings) and left intact for 1-7 days.
  Interventions: Device: Autologous Regeneration of Tissue (ART) device

INTERVENTIONS:
Device: Autologous Regeneration of Tissue (ART) device — This device will harvest hundreds of full-thickness columns of skin tissue (500 micrometer diameter) using single-needle, fluid-assisted harvesting technology.

SUMMARY:
The purpose of this research study is to learn about a new device, Autologous Regeneration of Tissue (ART), for collecting skin grafts from participant's own skin.

ELIGIBILITY:
Inclusion Criteria:

* Adults from 18 to 90 years of age.
* Patients that have a chronic wound in any area of the body defined as having been present for at least 30 days of duration.
* Able and willing to give consent for the study.

Exclusion Criteria:

* Pregnant women (Urine hCG test will be performed at baseline on women of child bearing potential).
* Adults unable to consent.
* Prisoners.
* Subjects requiring concurrent systemic antimicrobials during the study period for any infection.
* Subjects with leg lesions and clinically significant and unreconstructed peripheral arterial disease.
* Subjects who are receiving immunosuppressive agents, radiation therapy, or cytotoxic agents.
* Subjects who require treatment for a primary or metastatic malignancy (other than squamous or basal cell carcinoma of the skin).
* Subjects with other conditions considered by the investigator to be reasons for disqualification that may jeopardize subject safety or interfere with the objectives of the trial (e.g., acute illness or exacerbation of chronic illness, lack of motivation, history of poor compliance).

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2018-09-14 (Actual); Primary Completion 2024-03-19 (Actual); Study Completion 2024-03-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hadar Lev-Tov, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention Arm
Started | 22
Completed | 22
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Intervention Arm
Number analyzed (Participants) | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Change of Pain on Harvesting of Skin at Donor Site.
Description: Pain assessed using a Pain Visual Analog Scale (VAS) with a score ranging from 0 millimeters (no pain) to 100 millimeters (worst possible pain)
Time Frame: Baseline, Day 56
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Intervention Arm
Number analyzed (Participants) | 22
millimeters | 2.6 (5.9)

2. Primary Outcome: Time to Healing of Donor Sites
Description: At each weekly visit, the donor site will be assessed for healing based on clinical observation as measured by number of days from procedure.
Time Frame: Up to Day 56
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Intervention Arm
Number analyzed (Participants) | 22
Days | 24 (17)

3. Secondary Outcome: Wound Healing of Recipient Site
Description: At each weekly visit, the recipient area will be assessed for healing area percentage
Time Frame: Up to Day 56
Measure: Mean (Standard Deviation); unit: percentage of wound area healing
Arm/Group | Intervention Arm
Number analyzed (Participants) | 22
percentage of wound area healing | -3.6 (16.7)

4. Secondary Outcome: Histologic Evaluation
Description: As measured by tissue samples from biopsy
Time Frame: Up to Day 56
Population: This was an optional biopsy of the donor site at the final visit (approximately day 56). All participants opted to not participate in this optional procedure. Therefore, no data was collected.
Arm/Group | Intervention Arm
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 8 weeks.
Arm/Group | Intervention Arm
All-Cause Mortality (participants affected / at risk) | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22
Other Adverse Events (participants affected / at risk) | 11/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention Arm (N=22)
Bruising (Injury, poisoning and procedural complications) | 10 (10) — A grade 1 localized at the donor site.
Skin Infection (Infections and infestations) | 2 (2) — Participants that experienced a target wound Cellulitis.
Skin Infections (Infections and infestations) | 1 (1) — Participants that experienced cellulitis at the donor site.
Skin Infections (Infections and infestations) | 1 (1) — Participants that experienced contact dermatitis at the target wound.
Respiratory Infection (Infections and infestations) | 1 (1) — Participants that experienced COVID-19 symptoms.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2021-10-11): https://cdn.clinicaltrials.gov/large-docs/88/NCT03796988/Prot_001.pdf